CLINICAL TRIAL: NCT01923662
Title: Exploiting Selective Recruitment to Prolong Standing After SCI
Brief Title: A Neuroprosthesis for Prolonged Standing After SCI Using Multi-Contact Peripheral Nerve Electrodes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: B1039-R
Record Dates: First submitted 2013-08-07; First posted 2013-08-15 (Estimated); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injury; Paralysis; Tetraplegia; Paraplegia
Keywords: Paraplegia; Tetraplegia; Spinal Cord Injury; FES
MeSH Terms: conditions — Spinal Cord Injuries; Paralysis; Quadriplegia; Paraplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neuroprosthesis (Experimental): Eligible subjects will receive an implanted device (IRS-8 or IST-16) and surgically implanted electrodes to excite muscles that move paralyzed muscles. These electrodes are connected to the implanted stimulator that delivers electrical pulses to the nerves. These pulses cause the muscles to contract to perform functional movements or to exercise.
  Interventions: Device: IST-16 (16-Channel implanted stimulator-telemeter

INTERVENTIONS:
Device: IST-16 (16-Channel implanted stimulator-telemeter — Surgical implantation of IST-16 stimulator and electrodes to stimulate paralyzed muscles. Subjects will receive exercise and physical therapy with the implanted device. Functional training and laboratory assessments of clinical and technical performance will be conducted.

SUMMARY:
The purpose of this study is to improve the performance of neuroprosthesis for standing after SCI by developing and testing new advanced methods that use multiple contact peripheral nerve electrodes to slow the onset of fatigue and increase standing duration. The new advanced methods will take advantage of the ability of multiple-contact nerve cuff electrodes to selectively activate portions of a muscle that perform the same action. Alternating activation to multiple muscles (or parts of the same muscle) rather than continuously activation the entire muscle group constantly should allow them to rest and recover from fatiguing contractions. This should allow users to remain upright for longer periods of time to perform activities of daily living, reduce the risk of falls due to fatigue, and increase the potential of receiving the health benefits of standing.

DETAILED DESCRIPTION:
Neuroprostheses for standing after SCI currently rely on continuous activation of the hip and knee extensor muscles, which results in rapid fatigue and ultimately compromises elapsed standing time. The primary objective of this study is to improve the performance of neuroprostheses for standing by developing and implementing advanced stimulation paradigms that use multi-contact peripheral nerve electrodes to delay fatigue onset and prolong standing duration. The new stimulation paradigms will take advantage of the ability of multi-contact nerve cuff electrodes to selectively activate independent portions of a muscle, or independent muscles that perform the same action. Such a capability will allow one or more muscles (or parts of the same muscle) to rest while the others continue to contract to keep the knee extended and the user upright. Stimulation waveforms that alternate activation to multiple muscles performing the same function, rather than continuously activate the entire muscle group constantly, should allow muscles to rest and recover from fatiguing contractions.

In addition to these important clinical benefits, the project is also of high impact and significance because the methods to be developed will not be specific to any single electrode technology or stimulation system. Any clinical or therapeutic application that requires a sustained muscular contraction or the production of constant joint torques for prolonged periods of time will benefit from the successful completion of this project.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal maturity (age 21 and above), and ability to sign informed consent
* Paralysis resulting from neurological disorder such as low cervical/thoracic spinal cord injuries (C6-T12)
* Time post injury greater than six months to assure neurological and emotional stability
* Innervated and excitable lower extremity and lumbar trunk musculature
* Absence of acute or chronic psychological problems or chemical dependency
* Range of motion within normal limits, (full extension at the hip and knee, and ability to attain a neutral ankle position)
* Controlled spasticity and absence of hip flexion and adduction spasms
* Appropriate body habitus (BMI within normal range)
* Adequate social support and stability
* Willingness to comply with follow-up procedures.
* Full coverage of the acetabulum and minimal knee and ankle laxity

Exclusion Criteria:

* History of vestibular dysfunction, balance problems or spontaneous falls.
* Acute orthopaedic problems: severe scoliosis or joint dislocation, severe osteoporosis.
* Acute medical complication: cardiac abnormalities, skin breakdowns, uncontrolled seizures, or immunological, pulmonary/ renal/ circulatory compromise, auto-immune deficiencies, sepsis, active infection, dental caries.
* Diabetes
* Non-English speaking subjects
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04-11 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-03-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Triolo, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davis JA Jr, Triolo RJ, Uhlir J, Bieri C, Rohde L, Lissy D, Kukke S. Preliminary performance of a surgically implanted neuroprosthesis for standing and transfers--where do we stand? J Rehabil Res Dev. 2001 Nov-Dec;38(6):609-17. PMID 11767968
- [Background] Davis JA Jr, Triolo RJ, Uhlir JP, Bhadra N, Lissy DA, Nandurkar S, Marsolais EB. Surgical technique for installing an eight-channel neuroprosthesis for standing. Clin Orthop Relat Res. 2001 Apr;(385):237-52. doi: 10.1097/00003086-200104000-00035. PMID 11302320
- [Background] Fisher LE, Tyler DJ, Anderson JS, Triolo RJ. Chronic stability and selectivity of four-contact spiral nerve-cuff electrodes in stimulating the human femoral nerve. J Neural Eng. 2009 Aug;6(4):046010. doi: 10.1088/1741-2560/6/4/046010. Epub 2009 Jul 15. PMID 19602729
- [Background] Fisher LE, Miller ME, Bailey SN, Davis JA Jr, Anderson JS, Rhode L, Tyler DJ, Triolo RJ. Standing after spinal cord injury with four-contact nerve-cuff electrodes for quadriceps stimulation. IEEE Trans Neural Syst Rehabil Eng. 2008 Oct;16(5):473-8. doi: 10.1109/TNSRE.2008.2003390. PMID 18990650
- [Background] Uhlir JP, Triolo RJ, Kobetic R. The use of selective electrical stimulation of the quadriceps to improve standing function in paraplegia. IEEE Trans Rehabil Eng. 2000 Dec;8(4):514-22. doi: 10.1109/86.895955. PMID 11204043
- [Background] Chae J, Kilgore K, Triolo R, Creasey G. Functional neuromuscular stimulation in spinal cord injury. Phys Med Rehabil Clin N Am. 2000 Feb;11(1):209-26, x. PMID 10680166
- [Derived] Freeberg MJ, Pinault GCJ, Tyler DJ, Triolo RJ, Ansari R. Chronic nerve health following implantation of femoral nerve cuff electrodes. J Neuroeng Rehabil. 2020 Jul 14;17(1):95. doi: 10.1186/s12984-020-00720-3. PMID 32664972
- See also: APT Center is a VA Center of Excellence — http://www.aptcenter.research.va.gov
- See also: FES Center is VA Center of excellence — http://www.fescenter.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neuroprosthesis
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neuroprosthesis
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Average Standing Performance in Terms of Elapsed Standing Time for All Subjects.
Description: The investigators will assess standing performance in terms of elapsed standing time. The investigators will also collect data related to subjective impression of stability.
Time Frame: 12 months post-rehabilitation
Population: 5 participants with spinal cord injury with an implanted IST-16
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Neuroprosthesis
Number analyzed (Participants) | 5
Minutes | 32.6 (23.3)

2. Secondary Outcome: Percentage of Body Weight Distribution on the Legs While Standing With Stimulation.
Description: Determine the amount of weight on both legs during standing with stimulation.
Time Frame: 12 months post-rehabilitation
Population: 5 participants with spinal cord injury with an implanted IST-16
Measure: Mean (Standard Deviation); unit: % of body weight on lower extremity
Arm/Group | Neuroprosthesis
Number analyzed (Participants) | 5
% of body weight on lower extremity | 92.7 (.05)

ADVERSE EVENTS:
Time Frame: 8 years post implant
Arm/Group | Neuroprosthesis
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT01923662/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT01923662/ICF_001.pdf